CLINICAL TRIAL: NCT06536530
Title: MUDgame A Randomized Multi-Arm Controlled Experiment for Measuring the Benefits of an Exergame-based Intervention on Neuro-cognitive Functions in Adults Suffering From Depression
Brief Title: Benefits of Exergames on Neurocognitive Functions in Adults Suffering From Depression
Acronym: MUDGAME
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MAP Institute (Other)
Responsible Party: Principal Investigator, PhD Prof. Eloisa Ruiz-Marquez, Principal Investigator, MAP Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: z4s9q
Record Dates: First submitted 2024-07-23; First posted 2024-08-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: cognition; neuropsychology; neuroplasticity; event related potentials; exergames; video games
MeSH Terms: conditions — Depression | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: This project consists in a three-arms parallel-group randomized study to measure the benefits of exergames on cognition, in adults suffering from depression. Researchers will compare three different interventions (training with an exergame, which combines cognitive and physical stimulation, training with a cognitive game, and a wait-list condition), by randomizing participants to each group with equal probability.
Who Masked: Participant
Masking Description: This experiment is a single-blind design, where participants will be blind to the intervention, but researchers will not be blind to intervention allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exergame-Based Training (Experimental): Participants train with exergames (video games that include cognitive and physical training simultaneously), The training regime consists of 40-50 min sessions, two sessions per week, for a total of eight weeks of individual training.
  Interventions: Behavioral: Exergame-Based Training
- Cognitive-Based Training (Active Comparator): Participants will train only with cognitive video games. The training regime consists of 40-50 min sessions, two sessions per week, for a total of eight weeks of individual training.
  Interventions: Behavioral: Cognitive-Based Training
- Wait-List (Placebo Comparator): Participants will not train with any program and they will not assist to any specific session.
  Interventions: Behavioral: Wait-List

INTERVENTIONS:
Behavioral: Exergame-Based Training — 40-50 min sessions, two sessions per week, for a total of eight weeks.
  Arms: Exergame-Based Training
Behavioral: Cognitive-Based Training — 40-50 min sessions, two sessions per week, for a total of eight weeks.
  Arms: Cognitive-Based Training
Behavioral: Wait-List — Participants will not train with any program and they will not assist to any specific session or intervention
  Arms: Wait-List

SUMMARY:
The purpose of this study is to analyse the changes derived from exergames (videogames that include cognitive and physical stimulation simultaneously), in terms of cognitive functioning, psychomotor abilities, and its neural substrate, in adults suffering from depression.

DETAILED DESCRIPTION:
The experiment will consist in a randomized three-arms controlled study. After being informed about the study and potential risks, and given written informed consent, adult participants with depression will be randomly distributed into three experimental groups: an intervention group that will train with exergames, an active control group that will train only with cognitive games, and a passive control group or wait-list.

Cognitive Functions will be evaluated in three different moments: before the training intervention, after the intervention, and three months after finishing the training intervention.

Researchers will collect cognitive-behavioral and neural information (event-related potentials), and performing analysis of variance to compare the outcomes of the diverse groups at the three different time points, scientists will analyse the benefits of exergames on cognition.

ELIGIBILITY:
The inclusion and exclusion criteria for persons suffering from depression, will be validated by a professional (psychologist), through an interview and the use of reliable and valid psychological assessment tools.

Inclusion Criteria:

* Using the Beck Depression Inventory-Second Edition (BDI-II), a scored considered for inclusion criteria where depression (≥ 28 points on BDI-II), confirmed by psychological interview.
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* Participants suffering from depression with comorbidities (bipolar disorder, obsessive-compulsion disorder, neurological disorder, or traumatic brain injury) will be excluded.
* <20/60 vision with or without correction
* Inability to complete the activities
* Communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neuropsychological and Cognitive Functions (Executive Functions measured with the Wisconsin Card Sorting Test) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Executive functions (Wisconsin Card Sorting Test). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Baseline in Neuropsychological and Cognitive Functions (Memory will be measured with the tests Digit Spam Forward and Digit Spam Backward, from the Wechsler Memory Scale) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Memory (measured with the tests Digit Spam Forward and Digit Spam Backward, from the Wechsler Memory Scale). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Baseline in Neuropsychological and Cognitive Functions (Attention; sustained attention will be measured with the Sustained Attention to Response Task, SART) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Attention (measured with the Sustained Attention to Response Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Baseline in Neuropsychological and Cognitive Functions (Perception, visual perception will be measured with a classical Visual Search Task) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Perception (measured with a classical Visual Search Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Baseline in Neuropsychological and Cognitive Functions (Processing Speed, measured with a Simple Reaction Times Task) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Processing Speed (measured with a Simple Reaction Times Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Baseline in Neuropsychological and Cognitive Functions (Psychomotor functions, measured with the Salpêtrière Retardation Rating Scale) after eight weeks of training intervention or placebo condition. | Baseline and after eight weeks of training (Pre-assessment and Post-assessment)
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after eight weeks of training. Psychomotor functions (measured with the Salpetriere Retardation Rating Scale). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Executive functions measured with Wisconsin Card Sorting Test) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Executive functions (measured with Wisconsin Card Sorting Test). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Memory will be measured with the tests Digit Spam Forward and Digit Spam Backward, from the Wechsler Memory Scale) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Memory (measured with the tests Digit Spam Forward and Digit Spam Backward, from the Wechsler Memory Scale). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Attention; sustained attention will be measured with the Sustained Attention to Response Task) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Attention (measured with the Sustained Attention to Response Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Perception, visual perception will be measured with a classical Visual Search Task) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Perception (measured with a classical Visual Search Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Processing Speed, measured with a Simple Reaction Times Task) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Processing Speed (measured with a Simple Reaction Times Task). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).
Change from Post-assessment in Neuropsychological and Cognitive Functions (Psychomotor functions, measured with the Salpêtrière Retardation Rating Scale) after 3-month follow-up. | Three-month follow-up
  Researchers will use valid and realiable experimental tasks to measure the psychological functions after 3-month follow-up. Psychomotor functions (measured with the Salpetriere Retardation Rating Scale). The task mentioned here may be subject of modification. The measures include behavioral data (accuracy and reaction times) and neural data (event related potentials).
  (This test is going to be used as an experimental psychological task and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value in accuracy or reaction times).

SECONDARY OUTCOMES:
Change from Baseline in Placebo Effect measures (Motivation) after eight weeks of training. | Baseline and after eight weeks of training (Pre-assessment, Post-assessment)
  To measure the changes form baseline to the post-intervention, researchers will use to measure motivation a self-report 5-point Likert-type scale (1 = not motivated, to 5 = extremely motivated)
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).
Change from Baseline in Placebo Effect measures (Engagement) after eight weeks of training. | Baseline and after eight weeks of training (Pre-assessment, Post-assessment)
  To measure the changes form baseline to the post-intervention, researchers will use to measure engagement a self-report 5-point Likert-type scale (1 = not engaged, to 5 = extremely immersed).
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).
Change from Baseline in Placebo Effect measures (Expectations) after eight weeks of training. | Baseline and after eight weeks of training (Pre-assessment, Post-assessment)
  To measure the changes form baseline to the post-intervention, researchers will use to measure expectations, a self-report 5-point Likert-type (1 = the results will be much worse, 3 = there will not be any change, 5 = the results will be much better).
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).
Change from post-assessment in Placebo Effect measures (Motivation) after 3-month follow-up. | Three-month follow-up
  To measure the changes form post-test to the 3-month follow-up, researchers will use to measure motivation a self-report 5-point Likert-type scale (1 = not motivated, to 5 = extremely motivated)
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).
Change from post-assessment in Placebo Effect measures (Engagement) after 3-month follow-up. | Three-month follow-up
  To measure the changes form post-test to the 3-month follow-up, researchers will use to measure engagement a self-report 5-point Likert-type scale (1 = not engaged, to 5 = extremely immersed).
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).
Change from post-assessment in Placebo Effect measures (Expectations) after 3-month follow-up. | Three-month follow-up
  To measure the changes form post-test to the 3-month follow-up, researchers will use to measure expectations, a self-report 5-point Likert-type (1 = the results will be much worse, 3 = there will not be any change, 5 = the results will be much better).
  (This test is going to be used as a experimental self-report and it is not going to be used as a screening psychological tool, then, there are not cut-off values, a minimun or maximum value regarding the results).

IPD SHARING:
Plan to Share IPD: Yes
The available data will be individual participant data that underlie the results reported in the articles, after deidentification (text, tables, figures, and appendices), Study Protocol, Statistical Analysis Plan and Informed Consent Form.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available beginning 12 months and ending 3 years following articles publication.
URL: https://osf.io/ybdct/

REFERENCES:
- [Background] Ruiz-Marquez E. Neurophysiology of executive cognitive functions under depression. Explor Neurosci. 2025;4:100696. https://doi.org/10.37349/en.2025.100696
- [Background] Ruiz-Marquez E. Protocol for measuring the benefits of exergames on executive functions under depression through a randomized multi-arm controlled experiment. Explor Neurosci. 2024;3:564-83. https://doi.org/10.37349/en. 2024.00068
- [Background] Ruiz-Marquez, E. (2023). Protocol for measuring the benefits of exergames on executive functions under depression through a randomized multi-arm controlled experiment. Preprint. Open Science Framework.https://doi.org/10.31234/osf.io/m7s2t_v1
- [Background] Ruiz-Marquez, E. (2025). Neurophysiology of executive cognitive functions under depression. Preprint. Open Science Framework. https://doi.org/10.37349/en.2025.100696
- [Background] Ruiz-Marquez, E.,(2024). MUDgame. Measuring the Benefits of an Exergame-based intervention on Neuro-Cognitive Functions in adults suffering from Depression. A Randomized Multi-Arm Controlled Experiment. Project. Open Science Framework. https://doi.org/10.17605/OSF.IO/YBDCT
- [Background] Ruiz-Marquez, E. (2023). MUDgame. Measuring the Benefits of an Exergame-based intervention on Neuro-Cognitive Functions in adults suffering from Depression. A Randomized Multi-Arm Controlled Experiment. Preregistration. Open Science Framework. https://doi.org/10.17605/OSF.IO/Z4S9Q